CLINICAL TRIAL: NCT01303172
Title: A Randomised, Open-Label, Proof-of-Concept, Phase II Trial Comparing Gemcitabine With and Without IMM-101 in Advanced Pancreatic Cancer
Brief Title: A Trial Comparing Gemcitabine With and Without IMM-101 in Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Immodulon Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMM-101-002; IMAGE-1 (Other: Sponsor)
Record Dates: First submitted 2011-02-18; First posted 2011-02-24 (Estimated); Results first posted 2021-09-29 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Advanced Pancreatic Cancer
MeSH Terms: interventions — IMM-101; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine chemotherapy (Active Comparator): Patients in the control arm will receive normal standard of care - up to 12 cycles of Gemcitabine. Dosing of Gemcitabine is as per the normal prescribing information for pancreatic cancer.
  Interventions: Drug: Gemcitabine
- IMM-101 in addition to gemcitabine (Experimental): Patients in the experimental arm will receive IMM-101 in addition to the current standard of care, namely chemotherapy (Gemcitabine). The treatment regimen with IMM-101 will be every 2 weeks for the first 3 doses followed by a rest of 4 weeks then every 2 weeks for the next 3 doses followed by every 4 weeks thereafter.
  For patients in the active group, chemotherapy (Gemcitabine) will begin at least 14 days after first dose of IMM-101.
  Chemotherapy plus IMM-101 will be offered until intolerable toxicity or withdrawal from the study up to a maximum of 12 cycles (i.e. approximately 48 weeks).
  Patients who complete the Main Study and who provide informed consent are eligible to participate in a long term treatment Sub-Study (IMM-101-002A)
  Interventions: Biological: IMM-101

INTERVENTIONS:
Biological: IMM-101 — IMM-101 is a suspension of heat-killed whole cell M. obuense in borate-buffered saline.
  A single 0.1 mL intradermal injection of IMM-101 (10 mg/mL) will be administered every 2 weeks for the first 3 doses followed by a rest of 4 weeks then every 2 weeks for the next 3 doses followed by every 4 weeks thereafter.
  Chemotherapy plus IMM-101 will be offered until intolerable toxicity or withdrawal from the study up to a maximum of 12 cycles of gemcitabine.
  Other Names: Heat killed whole cell Mycobacterium obuense (M. obuense)
  Arms: IMM-101 in addition to gemcitabine
Drug: Gemcitabine — Gemcitabine will be administered intravenously at 1000 mg/m2 over 30 minutes once weekly for 3 consecutive weeks out of every 4 weeks.
  Chemotherapy will be offered until intolerable toxicity or withdrawal from the study up to a maximum of 12 cycles (i.e. approximately 48 weeks).
  Dosage reduction with each cycle or within each cycle may be applied based upon the grade of Gemcitabine-related toxicity experienced by the patient using centre's standard protocol.
  Other Names: Gemzar
  Arms: Gemcitabine chemotherapy

SUMMARY:
To compare, in patients with advanced pancreatic cancer, the effects of IMM-101 in combination with gemcitabine to gemcitabine alone on safety and tolerability (including QoL), clinical signs and symptoms of disease, selected markers of tumour burden and immunological status, and disease outcome.

DETAILED DESCRIPTION:
Patients in the IMM 101 treated group received an initial dose of IMM-101 followed by a maximum of 12 cycles of Gemcitabine (plus IMM-101); patients in the control group received Gemcitabine alone. All patients were to receive Gemcitabine once weekly for 3 consecutive weeks out of every 4 weeks. Patients in the IMM 101 treated group were to receive IMM 101 every 2 weeks for the first 3 doses, followed by a 4 week rest, then IMM-101 every 2 weeks for the next 3 doses. After this time, patients received doses every 4 weeks. Gemcitabine treatment began at least 14 days after the first dose of IMM-101 in the IMM 101 treated group.

Patients who completed the Main Study and who provided informed consent were eligible to participate in a long term treatment Sub-Study. All patients received IMM-101 in the open-label, single arm, Sub-Study irrespective of whether they had been randomised to Gemcitabine or Gemcitabine plus IMM-101 in the main study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female; aged ≥18 years.
* Histologically and/or cytologically confirmed inoperable ductal adenocarcinoma of the pancreas, including the mucinous variant. This will include locally advanced and metastatic disease (stage III/IV).
* Presence of measurable lesions in at least one site which have not been previously irradiated (bone lesions, ascites and pleural effusions are not considered as measurable), described as any of the following:

  * Any primary tumour with at least bi-dimensionally measurable disease.
  * a) Palpable lymph nodes; b) Deep seated lymph nodes.
  * Liver metastases measurable by computerised tomography (CT) scan.
  * Deep seated soft tissue lesions measurable by CT scan.
* World Health Organization (WHO) performance status of 0-2
* Serum creatinine <140 μmol/L
* White blood cell (WBC) count, including differential counts within the normal range or, if outside the normal range, considered by the Investigator not to be clinically significant.
* Life expectancy of >3 months from randomisation.
* Provided written informed consent to participate as shown by a signature and date on the patient's Informed Consent Form

Exclusion Criteria:

* Acinar cell carcinoma, neuroendocrine tumours, lymphomas or squamous cell carcinomas.
* Severe, active uncontrolled infection requiring systemic antibiotics, antiviral or antifungal treatments.
* Any previous chemotherapy treatment for pancreatic cancer.
* Eligible for resection of the pancreatic primary tumour but has either refused the operation or is considered to be medically unfit for the operation.
* Clinical or CT evidence of central nervous system (CNS) metastases.
* Any previous or concurrent malignancy, except adequately treated carcinoma in situ of the cervix, basal cell carcinoma of the skin and/or non-melanoma skin cancer, or if previous malignancy was more than 5 years earlier and there were no signs of recurrence.
* Any previous treatment with IMM-101 or related mycobacterial immunotherapy.
* Serum albumin < 26 g/L.
* C-reactive protein (CRP) > 70 mg/L.
* Radiotherapy in the 6 weeks prior to screening.
* Depot corticosteroids in the 6 weeks prior to screening.
* Chronic use of any systemic corticosteroids and/or immunosuppressant drugs within the 2-week period prior to the first administration of study drug.
* Female patient of child-bearing potential who is not, in the opinion of the Investigator, using an approved method of birth control.
* Female patient who were pregnant, breast feeding or planning a pregnancy during the course of the study. A pre-treatment serum pregnancy test measuring human chorionic gonadotrophin (hCG) had to be negative.
* Had been administered any investigational product e.g. drug, vaccine or device, in the 3 months prior to screening.
* Surgical or medical condition which, in the judgement of the Investigator, might interfere with the activity of IMM-101, or with the performance of this study.
* Any uncontrolled concomitant disease (e.g. unstable angina pectoris, congestive heart failure, myocardial infarction, arrhythmias, and uncontrolled severe hypertension) which, in the judgement of the Investigator, might interfere with the activity of IMM 101, or with the performance of this study.
* A history of serious adverse reaction or serious hypersensitivity to any drug.
* Known to have a history of human immunodeficiency virus (HIV) or syphilis, current symptomatic Hepatitis B or C. Testing is not required in the absence of clinical signs and symptoms suggestive of infection with HIV.
* Unable or unwilling to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angus Dalgleish, Professor, Principal Investigator — St George's, University of London
Locations (21):
- Cyprus Oncology Centre, Nicosia, Strovolos, Cyprus
- Ireland (2):
  - Adelaide, Meath & National Childrens Hospital,, Dublin
  - St Vicents University Hospital, Dublin
- Italy (4):
  - Azienda Ospedaliero-Universitaria di Bologna, Bologna
  - A.O. Santa Croce e Carle, Struttura Complessa di Oncologia Medica, Cuneo
  - Azienda Ospedaliera San Gerardo Struttura Complessa Oncologia Medica, Monza
  - AOU Maggiore della Carità, Novara
- Spain (6):
  - Medical Oncology Department, Central University Hospital of Asturias, Oviedo, Principality of Asturias
  - Hospital General de Alicante, Alicante
  - Hospital Gregorio Marañon, Madrid
  - Instituto Valenciano de Oncologia, Valencia
  - Department of Medical Oncology, Hospital Universitari La Fe,, Valencia
  - Hospital Miguel Servet, Zaragoza
- United Kingdom (8):
  - Airedale General Hospital, Skipton, West Yorkshire
  - Royal Blackburn Hospital, Blackburn
  - Bradford Royal Infirmary, Bradford
  - Velindre Cancer Centre, Cardiff
  - Ninewells Hospital,, Dundee
  - Mount Vernon Cancer Centre, London
  - The London Clinic Cancer Centre, London
  - Peterbrough City Hospital, Haematology/Oncology Dept,, Peterborough

REFERENCES:
- [Background] Dalgleish AG, Stebbing J, Adamson DJ, Arif SS, Bidoli P, Chang D, Cheeseman S, Diaz-Beveridge R, Fernandez-Martos C, Glynne-Jones R, Granetto C, Massuti B, McAdam K, McDermott R, Martin AJ, Papamichael D, Pazo-Cid R, Vieitez JM, Zaniboni A, Carroll KJ, Wagle S, Gaya A, Mudan SS. Randomised, open-label, phase II study of gemcitabine with and without IMM-101 for advanced pancreatic cancer. Br J Cancer. 2016 Sep 27;115(7):789-96. doi: 10.1038/bjc.2016.271. Epub 2016 Sep 6. PMID 27599039

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine Plus IMM-101: Patients in the experimental arm received IMM-101 in addition to Gemcitabine (Gem). The treatment regimen with IMM-101 was every 2 weeks for the first 3 doses followed by a rest of 4 weeks then every 2 weeks for the next 3 doses followed by every 4 weeks thereafter.
  For patients in the experimental group, GEM was initiated at least 14 days after first dose of IMM-101.
  GEM plus IMM-101 was offered until intolerable toxicity or withdrawal from the study up to a maximum of 12 cycles (i.e. approximately 48 weeks).
  IMM-101: IMM-101 is a suspension of heat-killed whole cell M. obuense in borate-buffered saline.
  A single 0.1 mL intradermal injection of IMM-101 (10 mg/mL)will be administered every 2 weeks for the first 3 doses followed by a rest of 4 weeks then every 2 weeks for the next 3 doses followed by every 4 weeks thereafter.
  Chemotherapy plus IMM-101 will be offered until intolerable toxicity or withdrawal from the study up to a maximum of 12 cycles of GEM.
  Patients who completed the Main Study and who provided informed consent were eligible to participate in a long term treatment Sub-Study where all patients received IMM-101.
- Gemcitabine Monotherapy: Patients in the control arm received normal standard of care - up to 12 cycles of Gemcitabine. Dosing of Gemcitabine was as per the normal prescribing information for pancreatic cancer.
  Gemcitabine was administered intravenously at 1000 mg/m2 over 30 minutes once weekly for 3 consecutive weeks out of every 4 weeks until intolerable toxicity or withdrawal from the study up to a maximum of 12 cycles (i.e. approximately 48 weeks).
  Dosage reduction with each cycle or within each cycle was applied based upon the grade of Gemcitabine-related toxicity experienced by the patient using centre's standard protocol.
  Patients who completed the Main Study and who provided informed consent were eligible to participate in a long term treatment Sub-Study where all patients received IMM-101.
Period: Overall Study
Arm/Group | Gemcitabine Plus IMM-101 | Gemcitabine Monotherapy
Started | 75 | 35
Completed | 12 | 1
Not Completed | 63 | 34
Not completed — Physician Decision | 9 | 6
Not completed — Adverse Event | 5 | 2
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Death | 20 | 7
Not completed — Lack of Efficacy | 25 | 17

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Gemcitabine plus IMM-101
- Control: Gemcitabine monotherapy
- Total: Total of all reporting groups
Arm/Group | Experimental | Control | Total
Number analyzed (Participants) | 75 | 35 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 16 | 44
  >=65 years | 47 | 19 | 66
Age, Continuous [Median (Full Range); unit: years] | 68 [45 to 88] | 66 [53 to 83] | 67 [45 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 14 | 51
  Male | 38 | 21 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 74 | 33 | 107
  Asian | 1 | 0 | 1
  Other | 0 | 1 | 1
  Unknown | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Cyprus | 3 | 3 | 6
  Ireland | 1 | 1 | 2
  United Kingdom | 25 | 9 | 34
  Italy | 14 | 9 | 23
  Spain | 32 | 13 | 45

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability.
Description: A clinically relevant deleterious effect of IMM-101 on safety and tolerability profiles was judged by:
  * Local and systemic toxicities.
  * Number, type and degree of toxicities as measured by the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) v4.0.
  Adverse events were collected from time of Informed Consent to 30 days post last dose of study medication IMM-101 does not appear to confer an incremental safety burden beyond that associated with chemotherapy and the disease itself. No new safety signals were identified from this study. The numbers of SAEs by preferred term were low, such that no trends could be inferred from these data and no significant SAEs attributable to IMM 101 were observed.
Time Frame: From time of Informed Consent to 30 days post last dose of study medication
Population: The safety analysis set included all randomised patients who received at least one dose of the study drug. One patient in the Gemcitabine plus IMM-101 group was withdrawn prior to administration of study treatment due to a worsening of his physical condition.
Measure: Number; unit: participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 74 | 35
participants
  With Treatment Emergent Adverse Events (TEAEs) | 73 | 35
  Withdrawn due to a TEAE | 4 | 0
  With TEAEs related to IMM-101 | 43 | 0
  With Treatment Emergent Serious Adverse Events (TESAEs) | 38 | 10
  With Treatment Emergent Serious Adverse Events (TESAEs) related to IMM-101 | 7 | 0

2. Secondary Outcome: Survival
Description: Overall and progression free survival
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year (or longer in the case of patients who entered the long term treatment sub-study, up to 5 years).
Population: The Intent To Treat analysis set included all randomised patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Experimental | Control
Number analyzed (Participants) | 75 | 35
Months
  Overall Survival | 6.7 [5.4 to 7.5] | 5.6 [3.2 to 7.2]
  Progression Free Survival | 4.1 [3.3 to 4.8] | 2.4 [2.1 to 4.0]

3. Secondary Outcome: Overall Response Rate (ORR).
Description: A clinically relevant improvement Overall Response Rate (ORR). Overall response rate was defined as the percentage of patients with a complete response or partial response as assessed by RECIST v1.1 criteria.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year (or longer in the case of patients who entered the long term treatment sub-study).
Population: The Intent To Treat analysis set included all randomised patients.
Measure: Number; unit: participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 75 | 35
participants
  Complete Response | 0 | 0
  Partial Response | 8 | 1

4. Secondary Outcome: Overall Survival in Metastatic Patients Only
Description: Overall and progression free survival in metastatic patients only
Time Frame: as for outcome 2
Population: The subgroup of patients with metastatic disease at baseline was the largest and accounted for 80.0% of patients in the ITT analysis set.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Experimental: IMM-101 plus Gemcitabine
Arm/Group | Experimental | Control
Number analyzed (Participants) | 64 | 28
Months | 7.0 [5.5 to 9.0] | 4.4 [2.8 to 6.5]
Statistical Analysis 1: Comparison: Experimental vs Control; The difference between the two treatment groups was tested with a two-sided log-rank test and a Cox regression model was used to estimate the hazard ratio (HR) and its 95% CI and associated p-value; Test type: Other; p = 0.011, Log Rank; Cox Proportional Hazard = 0.54, 95% CI 2-sided [0.33 to 0.87]

ADVERSE EVENTS:
Time Frame: Adverse event were collected and followed until resolution or for up to 30 days after the end of study/withdrawa
Description: It was the responsibility of the Investigator to document all AEs that occurred during the study. Adverse events were elicited by asking the patient a non-leading question, for example "Have you experienced or are you experiencing any new or changed symptoms since we last asked/since your last visit?" All AEs were followed until resolution or for up to 30 days after the end of study/withdrawal.
Arm/Group | Experimental | Control
All-Cause Mortality (participants affected / at risk) | 22/75 | 7/35
Serious Adverse Events (participants affected / at risk) | 36/75 | 10/35
Other Adverse Events (participants affected / at risk) | 73/75 | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=75) | Control (N=35)
Biliary sepsis (Infections and infestations) | 4 (6) | 0 (0)
Infection (Infections and infestations) | 3 (3) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (2)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (3) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection fungal (Infections and infestations) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 0 (0)
Ascites (Gastrointestinal disorders) | 3 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic duct stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 3 (3) | 2 (2)
Pyrexia (General disorders) | 4 (4) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
IVth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Nerve root compression (Nervous system disorders) | 1 (1) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulomonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arrhymia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=75) | Control (N=35)
Abdominal pain (Gastrointestinal disorders) | 35 (56) | 11 (22)
Diarrhoea (Gastrointestinal disorders) | 33 (65) | 14 (27)
Nausea (Gastrointestinal disorders) | 33 (59) | 13 (26)
Constipation (Gastrointestinal disorders) | 31 (42) | 11 (21)
Vomiting (Gastrointestinal disorders) | 22 (34) | 14 (19)
Stomatitis (Gastrointestinal disorders) | 8 (11) | 4 (8)
Ascites (Gastrointestinal disorders) | 7 (13) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 6 (7) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 9 (15) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 7 (9) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 6 (8) | 0 (0)
Gastrooesophageal reflux (Gastrointestinal disorders) | 6 (8) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 4 (6) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 4 (4) | 0 (0)
Asthenia (General disorders) | 34 (77) | 12 (46)
Fatigue (General disorders) | 19 (50) | 10 (24)
Pyrexia (General disorders) | 18 (30) | 2 (2)
Oedema peripheral (General disorders) | 12 (22) | 7 (9)
Mucosal inflammation (Gastrointestinal disorders) | 6 (8) | 1 (1)
Pain (General disorders) | 5 (6) | 2 (2)
Chills (General disorders) | 6 (7) | 0 (0)
Injection site reaction (General disorders) | 5 (8) | 0 (0)
Injection site pain (General disorders) | 4 (6) | 0 (0)
Oedema (General disorders) | 4 (6) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 33 (45) | 11 (24)
Vitamin D deficiency (Metabolism and nutrition disorders) | 7 (7) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 3 (5)
Anaemia (Blood and lymphatic system disorders) | 23 (40) | 9 (14)
Neutropenia (Blood and lymphatic system disorders) | 16 (48) | 10 (24)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (21) | 7 (13)
Leukopenia (Blood and lymphatic system disorders) | 4 (24) | 3 (9)
Weight decrased (Investigations) | 14 (17) | 1 (1)
Platelet count decrased (Investigations) | 7 (24) | 7 (14)
Alanine aminotransferase increased (Investigations) | 6 (15) | 2 (2)
Neutrophil count decreased (Investigations) | 5 (8) | 2 (3)
Blood bilirubin increased (Investigations) | 5 (12) | 1 (1)
WBC count deceased (Investigations) | 2 (7) | 4 (7)
Aspartate aminotransferase increased (Investigations) | 4 (11) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 4 (11) | 1 (2)
Haemoglobin deceased (Investigations) | 3 (10) | 2 (3)
Vitamin D decreased (Investigations) | 5 (6) | 0 (0)
Blood potassium decreased (Investigations) | 3 (10) | 2 (3)
Urinary tract infection (Infections and infestations) | 7 (10) | 3 (4)
Nasopharyngitis (Infections and infestations) | 5 (8) | 1 (3)
Respiratory tract infection (Infections and infestations) | 4 (6) | 0 (0)
Dysquesia (Nervous system disorders) | 13 (17) | 2 (2)
Lethargy (Nervous system disorders) | 9 (15) | 1 (2)
Dizziness (Nervous system disorders) | 8 (9) | 1 (1)
Headache (Nervous system disorders) | 8 (9) | 0 (0)
Parasthesia (Nervous system disorders) | 4 (4) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (24) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (9) | 2 (3)
Pruritis (Skin and subcutaneous tissue disorders) | 7 (8) | 2 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (6) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 6 (10) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (6) | 2 (3)
Insomnia (Psychiatric disorders) | 9 (9) | 3 (4)
Anxiety (Psychiatric disorders) | 9 (9) | 2 (4)
Depression (Psychiatric disorders) | 5 (6) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Jaundice (Hepatobiliary disorders) | 9 (10) | 1 (1)

LIMITATIONS AND CAVEATS:
This proof of concept study was not formally sized to test a specific pre-defined efficacy hypothesis. However, it has provided important insights into the potential for efficacy improvements with the use of IMM-101 in combination with chemotherapy in advanced pancreatic cancer.

Safety assessment based on AE & SAE profiles in each treatment arm had limitations as GEM is associated with frequent AEs and was given in both treatment arms. Thus, assessment of causality was difficult to interpret.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No